CLINICAL TRIAL: NCT02177214
Title: Prospective Study to Visualize Dynamesh ® IPOM Visible Mesh With MRI After Laparoscopic Intraperitoneal Ventral Hernia Repair.
Brief Title: Magnetic Resonance Imaging of Mesh Position After Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Head of the Department of Abdominal Surgery, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: IMAP STUDY; EuraHS (Registry Identifier: EuraHS)
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Hernia; Recurrence
MeSH Terms: conditions — Hernia; Recurrence | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ventral hernia: Adult patients scheduled for elective laparoscopic repair of ventral hernia, with inclusion of primary and incisional hernias. Visualization of the mesh surface observed with MRI scan at 3 weeks and 13 months after ventral hernia repair with a visible IPOM prosthesis (Dynamesh®)
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — Visualization of the mesh surface observed with MRI scan at 3 weeks and 13 months after ventral hernia repair with a visible IPOM prosthesis (Dynamesh®)

SUMMARY:
Purpose of the study is the visualization of the mesh and the determination of the mesh surface observed by MRI at 3 weeks and 13 months after ventral hernia repair with mesh visible IPOM (Dynamesh®). We want to prove that with this type of mesh it is possible to visualize the mesh position in vivo in a safe manner. This provides long-term benefit to early recognize possible recurrence caused by shifting or shrinking of the mesh and to provide early treatment.

DETAILED DESCRIPTION:
INTRODUCTION:

The repair of ventral hernias always goes along with a discussion about placing the optimal mesh, the optimum mesh position and the optimal fixation method of the mesh against the abdominal wall. There are a lot of meshes available of different materials, in different sizes and with different properties.

Penetrating fixation methods of the mesh have a strong positioning as result, but often at the cost of increased acute postoperative pain. Less or non-permanent (absorbable) fixation may decrease pain but should not risk a less stable mesh fixation ongoing with recurrence due to mesh shifting of mesh shrinkage.

It is indeed known that the majority of implanted meshes do shrink to an extent, which may be of disadvantage for the patient. This has already been demonstrated in several animal studies, but clinical information on the mesh shrinkage is rare and mostly a result from revised surgery.

All ordinary meshes for repair of abdominal hernia defects, based on polymeric textile, are invisible to conventional imaging techniques, inclusive "magnetic resonance imaging" (MRI). The IPOM mesh visible (Dynamesh®), developed by a unique method, contains an amount of iron particles, woven in the ordinary structure of the mesh, which allows an imaging in the MRI.

This study aims to visualize the implanted mesh in vivo by MRI. Furthermore, in cooperation with Dynamesh, we want to investigate the optimal concentration of iron particle resulting in optimal MRI.

PURPOSE Purpose of the study is the visualization of the mesh and the determination of the mesh surface observed by MRI at 3 weeks and 13 months after ventral hernia repair with mesh visible IPOM (Dynamesh®). We want to prove that with this type of mesh it is possible to visualize the mesh position in vivo in a safe manner. This provides long-term benefit to early recognize possible recurrence caused by shifting or shrinking of the mesh and to provide early treatment.

HERNIA REPAIR

* Introduction of the visible mesh IPOM (Dynamesh®) via laparoscopy and positioning against the abdominal wall with a minimum overlap with the hernia defect of at least 5 cm in all directions.
* The mesh will be fixed with absorbable staples, Secure Traps (Ethicon, Johnson & Johnson), in a double crown configuration. The staples are approximately 1.5 to 2 cm at distant from each other.
* All patients receive a standardized pain treatment protocol. Analgesics used will be checked. Visual analog scale (VAS) for pain will be measured at 4 hours, 8 hours, 12 hours, 16 hours, 20 hours and 24 hours post-operatively and every 12 hours thereafter until discharge of the patient.
* Pain medication after discharge will be monitored and checked with the patient at each consultation.

Clinical follow-up: clinical follow-up evaluations of patients at 1 and 13 months.

MRI measurement: post-operative scans and MRI analysis at 1 and 13 months.

DATA PROTECTION AND PRIVACY OF THE PATIENT All information about this study will be collected in EuraHS registry. The data will be entered into the EuraHS platform with a coded number, IMAP001, IMAP002, ...

LONG-TERM OUTCOME The ability to visualize the position of the intra-abdominal surgery mesh on the abdominal wall in a secure manner would be a huge step in abdominal wall surgery. It would give the surgeon the opportunity to quickly identify a possible loosening or moving or shrinking of the prosthesis and thus to prevent recurrence and other long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective laparoscopic repair of ventral hernia

Exclusion Criteria:

* - <18 years
* Lateral hernias (L1-L4), subxyphoidale hernias (M1) or suprapubicale hernias (M5).
* Emergency surgery (incarcerated hernia)
* Clean-contaminated or contaminated procedures
* ASA score> 4
* Pregnancy
* No patient Informed Consent
* Life expectancy of less than 2years
* Contra-indications for MRI examination, as of:
* Implanted electronic devices such as a pacemaker, neuro-stimulator, cochlear implant.
* Not MRI-compatible valves.
* Metal foreign bodies (depending on the location relative to the region to investigate).
* Large tattoos. Note: By default, the patient has to complete a questionnaire before the start of the study. This will be followed with the radiology nurse post-MRI.
* Claustrophobia, shortness of breath, tremor.
* In doubt, an internationally accepted list of items will be checked on the website www.mrisafety.com.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective laparoscopic repair of ventral hernia, with inclusion of primary and incisional hernias.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Visualization | 3 weeks
  Clear visualization of the MRI IPOM prosthesis 3 weeks postoperatively

SECONDARY OUTCOMES:
mesh surface | 13 month
  Calculation of mesh surface in comparison and% difference; visualization of IPOM prosthesis at 13 months postoperatively with MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muysoms FE, Novik B, Kyle-Leinhase I, Berrevoet F. Mesh fixation alternatives in laparoscopic ventral hernia repair. Surg Technol Int. 2012 Dec;22:125-32. PMID 23225589
- [Derived] Muysoms F, Beckers R, Kyle-Leinhase I. Prospective cohort study on mesh shrinkage measured with MRI after laparoscopic ventral hernia repair with an intraperitoneal iron oxide-loaded PVDF mesh. Surg Endosc. 2018 Jun;32(6):2822-2830. doi: 10.1007/s00464-017-5987-x. Epub 2017 Dec 21. PMID 29270800